CLINICAL TRIAL: NCT00369590
Title: Phase II Single Arm Trial of VEGF Trap in Patients With Recurrent Temozolomide-Resistant Malignant Gliomas
Brief Title: VEGF Trap in Treating Patients With Recurrent Malignant Gliomas That Did Not Respond to Temozolomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00677; NCI-2009-00677 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000495275; NABTC06-01 (Other: Adult Brain Tumor Consortium); NABTC-06-01 (Other: CTEP); U01CA062399 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-08

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Study Patients (Experimental): Patients receive VEGF Trap (ziv-aflibercept) IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study; laboratory biomarker analysis.
  Interventions: Biological: ziv-aflibercept; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap
Other: pharmacological study — correlative studies
Other: laboratory biomarker analysis — correlative studies

SUMMARY:
This phase II trial is studying how well VEGF Trap works in treating patients with recurrent malignant or anaplastic gliomas that did not respond to temozolomide. VEGF Trap may stop the growth of malignant or anaplastic gliomas by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the therapeutic efficacy of VEGF Trap in patients with temozolomide-resistant malignant gliomas at first recurrence as measured by 6-month progression-free survival (PFS).

II. Determine the safety profile of VEGF Trap in these patients.

SECONDARY OBJECTIVES:

I. Determine the efficacy of this regimen as measured by radiographic response, PFS, time to progression, and overall survival.

II. Characterize the single-dose and repeated-dose pharmacokinetic profiles of VEGF Trap in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to histology (glioblastoma vs anaplastic glioma).

Patients receive VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* International Normalized Ratio (INR) < = 1.5
* Platelet count => 100,000/mm³
* Hemoglobin => 10 g/dL (transfusion allowed)
* Serum glutamic oxaloacetic transaminase (SGOT)/Serum glutamic pyruvic transaminase (SGPT) < = 2 times upper limit of normal (ULN)
* Not pregnant or nursing
* Negative pregnancy test
* No previous Vascular endothelial growth factor (VEGF) Trap
* At least 4 weeks since chemotherapy, surgery, or open biopsy
* At least 2 weeks since vincristine
* At least 6 weeks since carmustine, lomustine, fotemustine, or radiation therapy
* At least 42 days since prior nitrosoureas
* At least 3 weeks since procarbazine
* No previous Gliadel wafers or bevacizumab
* Tumor did not respond to previous radiation therapy and temozolomide
* Karnofsky performance status (KPS) 60-100%
* Life expectancy = > 8 weeks
* White blood count (WBC) = >3,000/mm³
* Absolute neutrophil count = > 1,500/mm³
* Bilirubin < = 2 times ULN
* Creatinine < = 1.5 mg/dL OR creatinine clearance= > 60 mL/min
* Urine protein:creatinine ratio < = 1 OR 24-hour urine protein < = 500 mg/dL
* Fertile patients must use effective contraception prior to, during, and for = > 6 months after completion of study treatment
* No significant medical illnesses that, in the opinion of the investigator, cannot be adequately controlled with appropriate therapy or would preclude compliance with study treatment
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to other agents used in the study
* No history of any other cancer (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off of all therapy for that disease for = >3 years
* At least 7 days since prior noncytotoxic agents (e.g., interferon, tamoxifen, thalidomide, or isotretinoin [radiosensitizer does not count])
* At least 7 days since prior core biopsy
* At least 28 days since prior investigational agents
* No prior bevacizumab or vascular endothelial growth factor receptor inhibitors
* No concurrent full-dose anticoagulants (e.g., warfarin or low molecular-weight heparin)
* No clinically significant cardiovascular disease, including any of the following:

  * Cerebrovascular accident within the past 6 months
  * Uncontrolled hypertension, defined as blood pressure (BP) > 140/90 mm Hg or systolic BP > 180 mm Hg if diastolic BP < 90 mm Hg, on ≥ 2 repeated determinations on separate days within the past 3 months
  * Myocardial infarction, coronary artery bypass graft (CABG), or unstable angina pectoris within the past 6 months
  * New York Heart Association class III-IV congestive heart failure
  * No serious cardiac arrhythmia requiring medication
  * Clinically significant peripheral vascular disease within the past 6 months
  * Pulmonary embolism, deep vein thrombosis, or other thromboembolic event within the past 6 months
  * No evidence of bleeding diathesis or coagulopathy
* No more than 1 prior chemotherapy regimen (initial treatment and treatment for 1 relapse)
* Surgical resection for relapsed disease with no anticancer therapy instituted for up to 12 weeks followed by another surgical resection is considered 1 relapse
* If prior therapy for a grade 3 glioma was given, surgical diagnosis of a high-grade glioma is considered the first relapse
* Prior surgical, interstitial brachytherapy, or stereotactic radiosurgery not considered prior therapy
* If prior therapy included interstitial brachytherapy or stereotactic radiosurgery, must have confirmation of true progressive disease rather than radiation necrosis based upon either positron emission tomography (PET) scan, thallium scanning, Magnetic Resonance (MR) spectroscopy, or surgical documentation of disease
* Must show unequivocal radiographic evidence of tumor progression by MRI
* Recent resection of recurrent or progressive tumor allowed
* Residual disease not required
* Temozolomide-resistant recurrent glioblastoma is defined as tumor progression or tumor recurrence during or after treatment with temozolomide-based chemotherapy regimens
* Recovered from prior therapy
* No other disease that would obscure toxicity or dangerously alter drug metabolism
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situations that would limit compliance with study requirements
  * No serious or nonhealing wound, ulcer, or bone fracture
  * No history of intracerebral or intratumoral hemorrhage
  * No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
  * No significant traumatic injury within the past 28 days
* At least 28 days since prior cytotoxic therapy
* Histologically confirmed diagnosis of 1 of the following:

  * Intracranial glioblastoma or gliosarcoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified

    * NOTE: If original histology was grade 3 glioma, subsequent histological diagnosis of 1 of these diseases is allowed provided no prior diagnosis of grade 2 glioma
* At least 20 unstained slides OR 1 tissue block available from original diagnostic biopsy/surgery or from biopsy/surgery at recurrence
* Patients presenting at the time of first recurrence or relapse, defined as progression after initial therapy (i.e., radiotherapy +/- chemotherapy if that was used as initial therapy) are eligible
* No other concurrent investigational drugs
* No other concurrent investigational drugs
* No concurrent cytotoxic or noncytotoxic therapy, including chemotherapy, radiotherapy, hormonal therapy, or immunotherapy
* No concurrent major surgery
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent anticonvulsant therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-08; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John de Groot, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Background] de Groot JF, Lamborn KR, Chang SM, Gilbert MR, Cloughesy TF, Aldape K, Yao J, Jackson EF, Lieberman F, Robins HI, Mehta MP, Lassman AB, Deangelis LM, Yung WK, Chen A, Prados MD, Wen PY. Phase II study of aflibercept in recurrent malignant glioma: a North American Brain Tumor Consortium study. J Clin Oncol. 2011 Jul 1;29(19):2689-95. doi: 10.1200/JCO.2010.34.1636. Epub 2011 May 23. PMID 21606416
- [Derived] de Groot JF, Piao Y, Tran H, Gilbert M, Wu HK, Liu J, Bekele BN, Cloughesy T, Mehta M, Robins HI, Lassman A, DeAngelis L, Camphausen K, Chen A, Yung WK, Prados M, Wen PY, Heymach JV. Myeloid biomarkers associated with glioblastoma response to anti-VEGF therapy with aflibercept. Clin Cancer Res. 2011 Jul 15;17(14):4872-81. doi: 10.1158/1078-0432.CCR-11-0271. Epub 2011 Jun 1. PMID 21632852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (pts) were enrolled from Feb 2007 - Nov 2008. pts were from seven different cancer centers and were recruited from their outpatient cancer centers.
Groups:
- Arm I - Anaplastic Glioma; Arm 2 - Glioblastoma: Patients receive VEGF Trap (ziv-aflibercept) IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study; laboratory biomarker analysis.
  ziv-aflibercept: Given IV
  pharmacological study: correlative studies
  laboratory biomarker analysis: correlative studies
Period: Overall Study
Arm/Group | Arm I - Anaplastic Glioma | Arm 2 - Glioblastoma
Started | 16 | 42
Completed | 16 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 patients were anaplastic gliomas and 42 were glioblastomas all underwent central pathologic review
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Anaplastic Glioma | Arm 2 - Glioblastoma | Total
Number analyzed (Participants) | 16 | 42 | 58
Age, Continuous [Median (Full Range); unit: years] | 53 [26 to 70] | 55 [33 to 72] | 54 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 25 | 30
  Male | 11 | 17 | 28
Karnofsky Performance Status [Median (Full Range); unit: units on a scale] — The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment.
  100-80: Able to carry on normal activity and to work; No special care needed.
  70-50: Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed
  40-10: Unable to care for self; Requires equivalent of institutional or hospital care; diseases may be progressing rapidly.
  0: Dead
  units on a scale | 90 [60 to 100] | 90 [60 to 100] | 90 [60 to 100]
Pathology [Number; unit: participants]
  Glioblastoma | 0 | 39 | 39
  Gliosarcoma | 0 | 3 | 3
  Anaplastic astrocytoma | 12 | 0 | 12
  anaplastic oligodendroglioma | 3 | 0 | 3
  Anaplastic mixed oligoastrocytoma | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at 6 Months
Description: This design yields 85% power to detect a true 30% 6-month PFS rate, while maintaining .91 probability of rejecting for a true 15% 6-month PFS rate.
  pts had MRIs at screening and at the 3rd and 5th cycles then every 8 weeks until progression.
  Response determined by modified MacDonald Criteria Complete Response (CR): Complete disappearance of all measurable and evaluable disease, no new lesions. no steroids Partial Response (PR): Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable lesions. no new lesions. steroid dose no > than maximum dose used in first 8 weeks of treatment.
  Stable: Does not qualify for CR, PR, or progression steroid dose no > than maximum dose used in first 8 weeks of treatment.
  Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no increase) Clear clinical worsening.
Time Frame: 6 months
Population: pts not known to be progression free at time of the 6-month scan (24weeks) were considered to experienced treatment failure. If at least 10pts (24%) are progression-frree at 6months (GBM) the agent will be considered promising for futher study.
  The 3 pts in Arm 2 were treated at 2nd recurrence and were excluded from final efficacy analysis
Measure: Number; unit: percentage of participants
Arm/Group | Arm I - Anaplastic Glioma | Arm 2 - Glioblastoma
Number analyzed (Participants) | 16 | 39
percentage of participants | 25 | 7.7

2. Secondary Outcome: Response Rate Associated With VEGF Trap Therapy Defined as Proportions of Patients Experiencing Complete or Partial Response
Description: pts had MRIs at screening and at the 3rd and 5th cycles then every 8 weeks until progression. All responders were centrally reviewed for confirmation
  Response determined by modified MacDonald Criteria Complete Response (CR): Complete disappearance of all measurable and evaluable disease, no new lesions. no steroids Partial Response (PR): Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable lesions. no new lesions. steroid dose no > than maximum dose used in first 8 weeks of treatment.
  Stable: Does not qualify for CR, PR, or progression steroid dose no > than maximum dose used in first 8 weeks of treatment.
  Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no increase) Clear clinical worsening.
Time Frame: Up to 2 years
Population: The 3 pts in Arm 2 were treated at 2nd recurrence and were excluded from final efficacy analysis
Measure: Number; unit: participants
Arm/Group | Arm I - Anaplastic Glioma | Arm 2 - Glioblastoma
Number analyzed (Participants) | 16 | 39
participants
  Complete Response | 1 | 0
  Partial Response | 6 | 7

3. Primary Outcome: Safety Profile - Toxicities
Description: number of cycles patient was able to have before developing a toxicity that required removing the patient from treatment. Treatment: Aflibercept 4mg/kg intravenously on day 1 of every 14-day cycle - 2 week cycle.
Time Frame: Start to End of treatment 39 cycles or 1yr 7.5months (78 weeks)
Measure: Median (Full Range); unit: cycles
Arm/Group | Arm I - Anaplastic Glioma | Arm 2 - Glioblastoma
Number analyzed (Participants) | 16 | 42
cycles | 5 [1 to 39] | 3.5 [0 to 8]

4. Primary Outcome: Safety Profile - Events That Discontinued Treatment
Description: number of patients who experienced toxicity that led to being taken off treatment
Time Frame: Approximately 1 year (start of treatment - end of treatment)
Measure: Number; unit: participants
Arm/Group | Arm I - Anaplastic Glioma | Arm 2 - Glioblastoma
Number analyzed (Participants) | 16 | 42
participants | 8 | 6

5. Secondary Outcome: Progression Free Survival (PFS) Rate for Subjects With Radiographic Response
Description: pts with confirmed radiographic response and their rate of progression (PFS).
  Response determined by modified MacDonald Criteria Complete Response (CR): Complete disappearance of all measurable and evaluable disease, no new lesions. no steroids Partial Response (PR): Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable lesions. no new lesions. steroid dose no > than maximum dose used in first 8 weeks of treatment.
  Stable: Does not qualify for CR, PR, or progression steroid dose no > than maximum dose used in first 8 weeks of treatment.
  Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no increase) Clear clinical worsening.
Time Frame: up to 3 years
Population: Arm1 had total of 7 pts with response however, 2 pts stopped treatment early and were censored at 6 and 10 weeks.
  Arm 2 had total to 7 pts with response however 1 pt stopped treatment after 2 weeks but had a 4 week scan showing PR. - pt was censored.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm I - Anaplastic Glioma | Arm 2 - Glioblastoma
Number analyzed (Participants) | 5 | 6
weeks | 45 [24 to 134] | 23 [15 to 65]

6. Secondary Outcome: Overall Survival
Description: all patients alive as of the last contact were censored for survival on the basis of that contact date
Time Frame: 3 years
Population: The 3 pts in Arm 2 were treated at 2nd recurrence and were excluded from final efficacy analysis
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm I - Anaplastic Glioma | Arm 2 - Glioblastoma
Number analyzed (Participants) | 16 | 39
weeks | 55 [16 to 128] | 39 [3 to 150]

ADVERSE EVENTS:
Time Frame: adverse events were collected at baseline and at the end of each cycle until taken off treatment, approximately 1 yr
Groups:
- All Study Patients: Patients receive VEGF Trap (ziv-aflibercept) IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study; laboratory biomarker analysis.
  ziv-aflibercept: Given IV
  pharmacological study: correlative studies
  laboratory biomarker analysis: correlative studies
Arm/Group | All Study Patients
Serious Adverse Events (participants affected / at risk) | 3/58
Other Adverse Events (participants affected / at risk) | 35/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Patients (N=58)
ischemia cerebrovascular (Nervous system disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) — systemic hemorrhage
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Patients (N=58)
ataxia (Nervous system disorders) | 1 (1)
confusion (Psychiatric disorders) | 1 (1)
dysphaia (Nervous system disorders) | 1 (1)
fatigue (General disorders) | 3 (3)
palmar-plantar erythrodysesthesia syndrom (Skin and subcutaneous tissue disorders) | 1 (1) — hand-foot syndrome
headache (Nervous system disorders) | 1 (1)
hypertension (Vascular disorders) | 6 (6)
hyponatremia (Metabolism and nutrition disorders) | 2 (2)
hypophosphatejia (Metabolism and nutrition disorders) | 2 (2)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspartate aminotransferase increase (Investigations) | 1 (1)
lymphopenia (Investigations) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Neutrophil count decrease (Investigations) | 1 (1)
pain (General disorders) | 2 (2)
pericarditis (Cardiac disorders) | 1 (1)
proteinuria (Renal and urinary disorders) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
thromboembolic event (Vascular disorders) | 2 (2) — Thrombosis/embolism
wound complication (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less